CLINICAL TRIAL: NCT01771549
Title: Pilot Study of the Kinetics of High Sensitivity Troponin and Brain Natriuretic Peptide in Breast Cancer Chemotherapy With Adriamycin and Trastuzumab
Brief Title: Kinetics of Troponin and BNP in Breast Cancer Chemotherapy With Adriamycin and Trastuzumab
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph L. Blackshear, Principal Investigator, Mayo Clinic
Other Study IDs: 12-007541
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Adriamycin; Trastuzumab; Brain Natriuretic Peptide (BNP); Troponin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood 10 ml per draw, yielding 5 ml of serum. After testing, the remaining serum will be stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients with breast cancer beginning chemotherapy with a dose-dense regimen including adriamycin without concurrent trastuzumab.
- Group 2: Patients receiving trastuzumab in the adjuvant, neo-adjuvant, or metastatic setting in a regimen not containing simultaneous adriamycin therapy.

SUMMARY:
This pilot study involves very frequent monitoring of breast cancer patient blood levels of hs-cTnT Troponin and n-t-BNP (Brain Natriuretic Peptide) before and after initiation of chemotherapy with either adriamycin or trastuzumab in order to define the kinetics of both biomarkers during the first two cycles of chemotherapy. Cardiac troponins and BNP are frequently elevated after experimental chemotherapy in animal models. Their behavior in humans has been inconsistent, with occasional elevations seen, usually within 30 days of therapy. Assays for troponin with sensitivity into the pg/ml range have now been introduced. A majority of patients greater than age 50 have elevations above the detection limit, compared to only 1-3% with conventional troponin assays, and over 90% of diabetics have elevations above the detection limit. Moreover, augmented release of high sensitivity troponin is detected after exercise or rapid atrial pacing of durations of 10-15 minutes in patients with and without coronary artery disease. This improved sensitivity suggests the potential for detection and monitoring of cardiac damage after cancer chemotherapy. We hypothesized that this new generation of troponin assay would be associated with kinetic behavior suggesting ongoing cardiac damage with anthracycline therapy, and possibly also with trastuzumab.

DETAILED DESCRIPTION:
Collect blood samples in two groups of patients (n=10 per group) for amino-terminal brain natriuretic peptide (n-t-BNP) and high sensitivity cardiac troponin T (hs-cTnT):

* Group 1 (adriamycin) will consist of patients beginning clinically indicated chemotherapy for breast cancer with a dose-dense (every 2 week) regimen. including adriamycin (n=10).
* Group 2 will include patients who receive trastuzumab in the adjuvant or (neo) adjuvant setting, or in a metastatic setting in a regimen that does not include simultaneous adriamycin.

Blood samples for hs-cTNT and n-t-BNP will be obtained on days pre-treatment, and post-treatment days 1, 2, 3, 7, pre-cycle 2, and post-cycle 2 days 1,2,3 and 7. The interval for treatment is usually two weeks for adriamycin and three weeks for trastuzumab. We will identify frequency of detectible levels above the detection limit and above the baseline, peak values and area under the curve. Enrollment of up to 15 per group will be allowed to guarantee acquisition of 10 full sets of samples. Lab draw from chemotherapy ports will be allowed. We plan to store specimens for future analyses with more sensitive assays in development.

ELIGIBILITY:
Inclusion Criteria:

* Female adult patients aged 18+
* Group 1: beginning clinically- indicated chemotherapy for breast cancer with a dose-dense (every 2 weeks) regimen including adriamycin (n=10).
* Group 2: patients who receive trastuzumab in and adjuvant, (neo) adjuvant, or metastatic setting in a regimen that does not include simultaneous adriamycin.

Exclusion Criteria:

* Inability to return to the clinic for regular phlebotomy
* Baseline hemoglobin < 10 gm/dl
* Creatinine clearance < 60 ml/minute (this effects troponin clearance)
* Recent (< 3 months) cardiac surgery, myocardial infarction, unstable angina, or hospitalization for congestive heart failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic Florida female, adult patients from Hematology/Oncology Department undergoing clinically-indicated treatment for breast cancer which includes either, but not both, adriamycin or trastuzamab will be eligible to participate
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Area under the curve | one year
  Concentration-time plots from pre-treatment through days 1,2,3,7,and pre-cycle two

SECONDARY OUTCOMES:
Baseline to peak | 1 year
  The difference between the pretreatment value and the highest level on days 1,2,3 or 7

OTHER OUTCOMES:
Descriptive statistics | 1 year
  Descriptive statistics will be used to describe the quantitative values, and frequencies above and below the detection limit, time to peak, and amplitude of peak versus baseline values for both n-t-BNP and hs-cTnT.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Blackshear, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Result] Advani P, Hoyne J, Moreno-Aspita A, Dubin M, Brock S, Harlow C, Chumsri S, Suter T, Blackshear JL. High-Sensitivity Troponin T and NT-proBNP Kinetics in Breast Cancer Chemotherapy. Chemotherapy. 2017;62(6):334-338. doi: 10.1159/000477797. Epub 2017 Jul 14. PMID 28704807